CLINICAL TRIAL: NCT00474266
Title: Immunogenicity & Safety Study of GSK Biologicals' Meningococcal Vaccine GSK134612 When Co-Administered With GSK Biologicals' MMRV Vaccine (Priorix-Tetra™) in Healthy 12 to 23-Month-Old Children
Brief Title: Safety & Immunogenicity Study of Meningococcal Vaccine GSK134612 Given With Priorix-Tetra™ to 12-23 Month-Old Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109670; 2006-006580-23 (EudraCT Number)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infections, Meningococcal
Keywords: MMRV vaccine; co-administration; immunogenicity; meningococcal vaccine; conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — Priorix-Tetra vaccine

ARMS (4):
- Nimenrix + Priorix-Tetra Group (Experimental): Subjects received 1 dose of Nimenrix vaccine and 1 dose of Priorix-Tetra vaccine on Day 0 and a second dose of Priorix-Tetra vaccine on Day 84.
  Interventions: Biological: Meningococcal vaccine GSK134612 (Nimenrix); Biological: Priorix-Tetra
- Nimenrix Group (Experimental): Subjects received 1 dose of Nimenrix vaccine on Day 0 followed by 2 doses of Priorix-Tetra vaccine, respectively 42 and 84 days later.
  Interventions: Biological: Meningococcal vaccine GSK134612 (Nimenrix); Biological: Priorix-Tetra
- Priorix-Tetra Group (Active Comparator): Subjects received 1 dose of Priorix-Tetra vaccine on Day 0, 1 dose of Meningitec vaccine on Day 42 and a second dose of Priorix-Tetra vaccine on Day 84.
  Interventions: Biological: Priorix-Tetra; Biological: Meningitec
- Meningitec Group (Active Comparator): Subjects received 1 dose of Meningitec vaccine on Day 0 followed by 2 doses of Priorix-Tetra vaccine, respectively 42 and 84 days later.
  Interventions: Biological: Priorix-Tetra; Biological: Meningitec

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 (Nimenrix) — Single dose intramuscular injection
  Arms: Nimenrix + Priorix-Tetra Group; Nimenrix Group
Biological: Priorix-Tetra — 2-dose subcutaneous injection
Biological: Meningitec — Single dose intramuscular injection
  Arms: Meningitec Group; Priorix-Tetra Group

SUMMARY:
The purpose of this study is to demonstrate, in 12-23 month old children, the non-inferiority of the meningococcal vaccine 134612 given with Priorix-Tetra.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Open multicentre study with 4 treatment groups. Two groups will receive the 134612 vaccine with Priorix-Tetra either at the same or different visits followed by a second Priorix-Tetra vaccination at 84 days.

Two control groups will receive Priorix-Tetra and Meningitec at different visits followed by a second Priorix-Tetra vaccination at 84 days.

For all subjects, two blood samples will be taken: prior to and 42 days after the first vaccination. In a subset (30% of subjects in Groups A en C) from selected study centres: additional sample 42 days after second Priorix-Tetra dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 23 months of age at the time of the vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of parents' or legal guardians' knowledge.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month before and 42 days after the first dose of vaccine(s).
* Previous vaccination with meningococcal vaccine of serogroup A, C W and/or Y.
* History of meningococcal disease.
* Previous vaccination against measles, mumps, rubella, and/or varicella.
* History of measles, mumps, rubella and/or varicella.
* Known exposure to measles, mumps, rubella, varicella or zoster within 30 days prior to vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including neomycin.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2007-06-05 (Actual); Primary Completion 2008-02-26 (Actual); Study Completion 2008-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=248

REFERENCES:
- [Background] Vesikari T, Karvonen A, Bianco V, Van der Wielen M, Miller J. Tetravalent meningococcal serogroups A, C, W-135 and Y conjugate vaccine is well tolerated and immunogenic when co-administered with measles-mumps-rubella-varicella vaccine during the second year of life: An open, randomized controlled trial. Vaccine. 2011 Jun 6;29(25):4274-84. doi: 10.1016/j.vaccine.2011.03.043. Epub 2011 Apr 6. PMID 21443965
- [Background] Vesikari T, Forsten A, Bianco V, Van der Wielen M, Miller JM. Immunogenicity, Safety and Antibody Persistence of a Booster Dose of Quadrivalent Meningococcal ACWY-tetanus Toxoid Conjugate Vaccine Compared with Monovalent Meningococcal Serogroup C Vaccine Administered Four Years After Primary Vaccination Using the Same Vaccines. Pediatr Infect Dis J. 2015 Dec;34(12):e298-307. doi: 10.1097/INF.0000000000000897. PMID 26780033
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix + Priorix-Tetra Group: Subjects received 1 dose of Nimenrix™ vaccine and 1 dose of Priorix-Tetra™ vaccine on Day 0 and a second dose of Priorix-Tetra™ vaccine on Day 84.
- Nimenrix Group: Subjects received 1 dose of Nimenrix™ vaccine on Day 0 followed by 2 doses of Priorix-Tetra™ vaccine, respectively 42 and 84 days later.
- Priorix-Tetra Group: Subjects received 1 dose of Priorix-Tetra™ vaccine on Day 0, 1 dose of Meningitec™ vaccine on Day 42 and a second dose of Priorix-Tetra™ vaccine on Day 84.
- Meningitec Group: Subjects received 1 dose of Meningitec™ vaccine on Day 0 followed by 2 doses of Priorix-Tetra™ vaccine, respectively 42 and 84 days later.
Period: Overall Study
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Started | 375 | 374 | 126 | 125
Completed | 368 | 354 | 122 | 118
Not Completed | 7 | 20 | 4 | 7
Not completed — Withdrawal by Subject | 7 | 20 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group | Total
Number analyzed (Participants) | 375 | 374 | 126 | 125 | 1000
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.7 (1.5) | 14.6 (1.49) | 14.6 (1.41) | 14.4 (1.47) | 14.61 (1.48)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 180 | 174 | 68 | 60 | 482
  Male | 195 | 200 | 58 | 65 | 518
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/ European heritage, n (%) | 369 | 372 | 123 | 123 | 987
  Other | 4 | 2 | 2 | 2 | 10
  White - Arabic / North African heritage | 2 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With rSBA-MenC, rSBA-MenA, rSBA-MenW-135, rSBA-MenY Titers Greater Than or Equal to (≥) the Cut-off Values
Description: The cut-off values for the rSBA titers were ≥ 1:8. The analysis was performed only on subjects receiving meningitis vaccination (Nimenrix) at Day 0.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Meningitec Group
Number analyzed (Participants) | 360 | 354 | 121
Participants
  rSBA-MenA, D42: number analyzed (Participants) | 360 | 354 | 51
  rSBA-MenA, D42 | 360 | 353 | 23
  rSBA-MenC, D42: number analyzed (Participants) | 357 | 354 | 121
  rSBA-MenC, D42 | 357 | 353 | 118
  rSBA-MenW-135, D42: number analyzed (Participants) | 360 | 354 | 58
  rSBA-MenW-135, D42 | 360 | 354 | 29
  rSBA-MenY, D42: number analyzed (Participants) | 359 | 354 | 59
  rSBA-MenY, D42 | 359 | 354 | 32
Statistical Analysis 1: Comparison: Nimenrix Group vs Meningitec Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage = 2.2, 95% CI 2-sided [0.29 to 6.78]
Statistical Analysis 2: Comparison: Nimenrix + Priorix-Tetra Group vs Nimenrix Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥ -10%; Difference in percentage = 0.28, 95% CI 2-sided [-0.78 to 1.58]
Statistical Analysis 3: Comparison: Nimenrix + Priorix-Tetra Group vs Nimenrix Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥ -10%; Difference in percentage = 0.28, 95% CI 2-sided [-0.79 to 1.58]
Statistical Analysis 4: Comparison: Nimenrix + Priorix-Tetra Group vs Nimenrix Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-1.06 to 1.07]

2. Primary Outcome: Number of Subjects With Anti-measles Antibody Concentrations ≥ the Cut-off Values
Description: The cut-off values for anti-measles antibody concentrations were ≥ 150 milli-international units per milliliter (mIU/mL).
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 361 | 354 | 118 | 120
Participants | 361 | 0 | 118 | 0
Statistical Analysis 1: Comparison: Nimenrix + Priorix-Tetra Group vs Priorix-Tetra Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-1.06 to 3.17]

3. Primary Outcome: Number of Subjects With Anti-mumps Antibody Concentrations ≥ the Cut-off Values
Description: The cut-off values for anti-mumps antibody concentrations were ≥ 231 units per milliliter (U/mL).
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 349 | 354 | 116 | 120
Participants | 306 | 0 | 97 | 0
Statistical Analysis 1: Comparison: Nimenrix + Priorix-Tetra Group vs Priorix-Tetra Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage = 4.06, 95% CI 2-sided [-2.82 to 12.46]

4. Primary Outcome: Number of Subjects With Anti-rubella Antibody Concentrations ≥ the Cut-off Values.
Description: The cut-off values for anti-rubella antibody concentrations were ≥ 4 international units per milliliter (IU/mL).
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 361 | 354 | 118 | 120
Participants | 361 | 1 | 118 | 1
Statistical Analysis 1: Comparison: Nimenrix + Priorix-Tetra Group vs Priorix-Tetra Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-1.06 to 3.18]

5. Primary Outcome: Number of Subjects With Anti-varicella Antibody Concentrations ≥ the Cut-off Values
Description: The cut-off values for anti-varicella antibody concentrations were ≥ 1:4.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 333 | 335 | 111 | 116
Participants | 326 | 6 | 105 | 2
Statistical Analysis 1: Comparison: Nimenrix + Priorix-Tetra Group vs Priorix-Tetra Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage = 3.36, 95% CI 2-sided [-0.28 to 9.5]

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off values for the rSBA titers were ≥ 1:8 and ≥ 1:128 respectively. At pre-vaccination for all groups, half of the subjects were sera tested for rSBA-MenC while the other half was tested for rSBA-MenA, rSBA-MenW-135 and rSBA-MenY. At Post vaccination I (Day 42), all subjects from Nimenrix + Priorix-Tetra and Nimenrix groups were sera tested for each rSBA. For Meningitec and Priorix-Tetra groups, all subjects were tested for rSBA-MenC while half of subjects were tested for rSBA-MenA, rSBA-MenW-135 and rSBA-MenY.
Time Frame: Prior to vaccination (Day 0) and after the first vaccination dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 360 | 354 | 117 | 121
Participants
  rSBA-MenA ≥ 1:8, D0: number analyzed (Participants) | 158 | 171 | 53 | 53
  rSBA-MenA ≥ 1:8, D0 | 57 | 77 | 24 | 18
  rSBA-MenA ≥ 1:128, D0: number analyzed (Participants) | 158 | 171 | 53 | 53
  rSBA-MenA ≥ 1:128, D0 | 32 | 50 | 18 | 10
  rSBA-MenA ≥ 1:128, D42: number analyzed (Participants) | 360 | 354 | 55 | 51
  rSBA-MenA ≥ 1:128, D42 | 359 | 353 | 22 | 17
  rSBA-MenC ≥ 1:8, D0: number analyzed (Participants) | 178 | 174 | 60 | 60
  rSBA-MenC ≥ 1:8, D0 | 48 | 47 | 16 | 13
  rSBA-MenC ≥ 1:128, D0: number analyzed (Participants) | 178 | 174 | 60 | 60
  rSBA-MenC ≥ 1:128, D0 | 19 | 22 | 4 | 4
  rSBA-MenC ≥ 1:128, D42: number analyzed (Participants) | 357 | 354 | 117 | 121
  rSBA-MenC ≥ 1:128, D42 | 337 | 339 | 13 | 85
  rSBA-MenW-135 ≥ 1:8, D0: number analyzed (Participants) | 177 | 177 | 60 | 61
  rSBA-MenW-135 ≥ 1:8, D0 | 76 | 81 | 29 | 30
  rSBA-MenW-135 ≥ 1:128, D0: number analyzed (Participants) | 177 | 177 | 60 | 61
  rSBA-MenW-135 ≥ 1:128, D0 | 30 | 28 | 14 | 12
  rSBA-MenW-135 ≥ 1:128, D42: number analyzed (Participants) | 360 | 354 | 58 | 58
  rSBA-MenW-135 ≥ 1:128, D42 | 360 | 352 | 16 | 15
  rSBA-MenY ≥ 1:8, D0: number analyzed (Participants) | 179 | 181 | 60 | 62
  rSBA-MenY ≥ 1:8, D0 | 103 | 112 | 41 | 34
  rSBA-MenY ≥ 1:128, D0: number analyzed (Participants) | 179 | 181 | 60 | 62
  rSBA-MenY ≥ 1:128, D0 | 75 | 79 | 30 | 23
  rSBA-MenY ≥ 1:128, D42: number analyzed (Participants) | 359 | 354 | 58 | 59
  rSBA-MenY ≥ 1:128, D42 | 358 | 353 | 30 | 21

7. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Antibody titers were expressed as geometric mean titers (GMTs). At pre-vaccination for all groups, half of the subjects were sera tested for rSBA-MenC while the other half were tested for rSBA-MenA, rSBA-MenW-135 and rSBA-MenY. At Post vaccination I (Day 42), all subjects from Nimenrix + Priorix-Tetra and Nimenrix groups were sera tested for each rSBA. For Meningitec and Priorix-Tetra groups, all subjects were tested for rSBA-MenC while half of subjects were tested for rSBA-MenA, rSBA-MenW-135 and rSBA-MenY.
Time Frame: Prior to first vaccine dose (Day 0) and 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 360 | 354 | 117 | 121
Titer
  rSBA-MenA, D0: number analyzed (Participants) | 158 | 171 | 53 | 53
  rSBA-MenA, D0 | 14.6 [10.9 to 19.4] | 22.8 [16.8 to 31] | 24.4 [13.7 to 43.4] | 14.3 [8.5 to 24]
  rSBA-MenA, D42: number analyzed (Participants) | 360 | 354 | 55 | 51
  rSBA-MenA, D42 | 2085.9 [1905.3 to 2283.6] | 2205 [2007.8 to 2421.6] | 33.1 [19.1 to 57.4] | 24.3 [13.4 to 44.1]
  rSBA-MenC, D0: number analyzed (Participants) | 178 | 174 | 60 | 60
  rSBA-MenC, D0 | 9.2 [7.4 to 11.4] | 10 [7.8 to 12.6] | 8.5 [6 to 12.2] | 7.6 [5.5 to 10.6]
  rSBA-MenC, D42: number analyzed (Participants) | 357 | 354 | 117 | 121
  rSBA-MenC, D42 | 519 [470.9 to 571.9] | 477.6 [437.3 to 521.6] | 11.2 [8.3 to 15.2] | 212.3 [170 to 265.2]
  rSBA-MenW-135, D0: number analyzed (Participants) | 177 | 177 | 60 | 61
  rSBA-MenW-135, D0 | 16.2 [12.6 to 20.7] | 16.7 [13.1 to 21.4] | 21.9 [13.5 to 35.4] | 20.8 [13.1 to 33.2]
  rSBA-MenW-135, D42: number analyzed (Participants) | 360 | 354 | 58 | 58
  rSBA-MenW-135, D42 | 2055.8 [1871 to 2258.9] | 2681.7 [2453.1 to 2931.6] | 25.6 [15.6 to 42.1] | 25.1 [14.6 to 43.1]
  rSBA-MenY, D0: number analyzed (Participants) | 179 | 181 | 60 | 62
  rSBA-MenY, D0 | 41.4 [30.2 to 56.6] | 50.1 [36.7 to 68.2] | 71 [40.9 to 123.2] | 31.7 [18.9 to 53.2]
  rSBA-MenY, D42: number analyzed (Participants) | 359 | 354 | 58 | 59
  rSBA-MenY, D42 | 2282.4 [2051.3 to 2539.5] | 2729.4 [2472.7 to 3012.8] | 70 [39.3 to 124.7] | 31.4 [18.4 to 53.6]

8. Secondary Outcome: Anti-PSA (Anti-polysaccharide A), Anti-PSC, Anti-PSW-135 and Anti-PSY Antibodies Concentrations ≥ the Cut-off Values
Description: Anti-PS antibody concentrations were given as geometric mean concentrations (GMCs) and expressed as microgram per milliliter (μg/mL). At pre-vaccination (Day 0) and Post-vaccination I (Day 42), a quarter of the subjects were tested for anti-PSC and another quarter for anti-PSA, anti-PSW-135 and anti-PSY.
Time Frame: Prior to the first vaccine dose (Day 0) and 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 90 | 93 | 30 | 31
μg/mL
  Anti-PSA, D0: number analyzed (Participants) | 90 | 93 | 29 | 31
  Anti-PSA, D0 | 0.17 [0.15 to 0.19] | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.18] | 0.16 [0.14 to 0.17]
  Anti-PSA, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSA, D42 | 28.74 [24.01 to 34.4] | 15.71 [12.91 to 19.12] | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.17]
  Anti-PSC, D0: number analyzed (Participants) | 89 | 90 | 30 | 30
  Anti-PSC, D0 | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15]
  Anti-PSC, D42: number analyzed (Participants) | 89 | 87 | 29 | 29
  Anti-PSC, D42 | 9.26 [7.73 to 11.1] | 7.44 [6.43 to 8.6] | 0.15 [0.15 to 0.15] | 4.89 [3.69 to 6.47]
  Anti-PSW-135, D0: number analyzed (Participants) | 90 | 92 | 29 | 31
  Anti-PSW-135, D0 | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.18] | 0.15 [0.15 to 0.15]
  Anti-PSW-135, D42: number analyzed (Participants) | 90 | 92 | 29 | 31
  Anti-PSW-135, D42 | 6.5 [5.52 to 7.65] | 4.5 [3.77 to 5.37] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.15]
  Anti-PSY, D0: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSY, D0 | 0.15 [0.15 to 0.15] | 0.16 [0.15 to 0.16] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15]
  Anti-PSY, D42: number analyzed (Participants) | 89 | 93 | 29 | 31
  Anti-PSY, D42 | 8.56 [7.26 to 10.11] | 6.37 [5.13 to 7.92] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.15]

9. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibodies Concentrations ≥ the Cut-off Values
Description: The cut-off values for anti-PS antibody concentrations were ≥ 0.3 μg/mL and ≥ 2.0 μg/mL respectively. At pre-vaccination (Day 0) and Post-vaccination I (Day 42), a quarter of the subjects were tested for anti-PSC and another quarter for anti-PSA, anti-PSW-135 and anti-PSY.
Time Frame: Prior to first vaccine dose (Day 0) and 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 90 | 93 | 30 | 31
Participants
  Anti-PSA ≥ 0.3 μg/mL, D0: number analyzed (Participants) | 90 | 93 | 29 | 31
  Anti-PSA ≥ 0.3 μg/mL, D0 | 6 | 1 | 1 | 1
  Anti-PSA ≥ 0.3 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSA ≥ 0.3 μg/mL, D42 | 90 | 89 | 2 | 1
  Anti-PSA ≥ 2 μg/mL, D0: number analyzed (Participants) | 90 | 93 | 29 | 31
  Anti-PSA ≥ 2 μg/mL, D0 | 0 | 0 | 0 | 0
  Anti-PSA ≥ 2 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSA ≥ 2 μg/mL, D42 | 90 | 88 | 0 | 0
  Anti-PSC ≥ 0.3 μg/mL, D0: number analyzed (Participants) | 89 | 90 | 30 | 30
  Anti-PSC ≥ 0.3 μg/mL, D0 | 0 | 0 | 0 | 0
  Anti-PSC ≥ 0.3 μg/mL, D42: number analyzed (Participants) | 89 | 87 | 29 | 29
  Anti-PSC ≥ 0.3 μg/mL, D42 | 89 | 87 | 0 | 29
  Anti-PSC ≥ 2 μg/mL, D0: number analyzed (Participants) | 89 | 90 | 30 | 30
  Anti-PSC ≥ 2 μg/mL, D0 | 0 | 0 | 0 | 0
  Anti-PSC ≥ 2 μg/mL, D42: number analyzed (Participants) | 89 | 87 | 29 | 29
  Anti-PSC ≥ 2 μg/mL, D42 | 85 | 85 | 0 | 26
  Anti-PSW-135 ≥ 0.3 μg/mL, D0: number analyzed (Participants) | 90 | 92 | 29 | 31
  Anti-PSW-135 ≥ 0.3 μg/mL, D0 | 4 | 2 | 1 | 0
  Anti-PSW-135 ≥ 0.3 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSW-135 ≥ 0.3 μg/mL, D42 | 90 | 89 | 1 | 0
  Anti-PSW-135 ≥ 2 μg/mL, D0: number analyzed (Participants) | 90 | 92 | 29 | 31
  Anti-PSW-135 ≥ 2 μg/mL, D0 | 0 | 0 | 0 | 0
  Anti-PSW-135 ≥ 2 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSW-135 ≥ 2 μg/mL, D42 | 82 | 80 | 0 | 0
  Anti-PSY ≥ 0.3 μg/mL, D0: number analyzed (Participants) | 89 | 93 | 29 | 31
  Anti-PSY ≥ 0.3 μg/mL, D0 | 0 | 4 | 0 | 0
  Anti-PSY ≥ 0.3 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSY ≥ 0.3 μg/mL, D42 | 90 | 89 | 1 | 0
  Anti-PSY ≥ 2 μg/mL, D0: number analyzed (Participants) | 89 | 93 | 29 | 31
  Anti-PSY ≥ 2 μg/mL, D0 | 0 | 0 | 0 | 0
  Anti-PSY ≥ 2 μg/mL, D42: number analyzed (Participants) | 90 | 90 | 29 | 30
  Anti-PSY ≥ 2 μg/mL, D42 | 87 | 79 | 0 | 0

10. Secondary Outcome: Number of Subjects With hSBA-MenA (Meningococcal Polysaccharide A Serum Bactericidal Antibodies Using Human Complement), hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off values for hSBA antibody titers were ≥ 1:4 and ≥ 1:8 for Nimenrix + Priorix-Tetra group, Nimenrix group, Meningitec group and Pooled group (Nimenrix + Priorix-Tetra and Nimenrix groups), respectively. The analysis was performed only on subjects receiving meningitis vaccination (Nimenrix) at Day 0.
Time Frame: Prior to first vaccine dose (Day 0) and 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Group: Subjects from Nimenrix + Priorix-Tetra Group and subjects from Nimenrix Group
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Meningitec Group | Pooled Group
Number analyzed (Participants) | 359 | 363 | 123 | 722
Participants
  hSBA-MenA ≥1:4, D0: number analyzed (Participants) | 357 | 356 | 122 | 713
  hSBA-MenA ≥1:4, D0 | 14 | 8 | 2 | 22
  hSBA-MenA ≥1:4, D42: number analyzed (Participants) | 348 | 338 | 117 | 686
  hSBA-MenA ≥1:4, D42 | 305 | 273 | 1 | 578
  hSBA-MenA ≥1:8, D0: number analyzed (Participants) | 357 | 356 | 122 | 713
  hSBA-MenA ≥1:8, D0 | 7 | 7 | 1 | 14
  hSBA-MenA ≥1:8, D42: number analyzed (Participants) | 348 | 338 | 123 | 686
  hSBA-MenA ≥1:8, D42 | 292 | 261 | 1 | 553
  hSBA-MenC ≥1:4, D0: number analyzed (Participants) | 359 | 363 | 122 | 722
  hSBA-MenC ≥1:4, D0 | 1 | 3 | 1 | 4
  hSBA-MenC ≥1:4, D42: number analyzed (Participants) | 346 | 341 | 116 | 687
  hSBA-MenC ≥1:4, D42 | 339 | 339 | 95 | 677
  hSBA-MenC ≥1:8, D0: number analyzed (Participants) | 359 | 363 | 122 | 722
  hSBA-MenC ≥1:8, D0 | 1 | 3 | 1 | 4
  hSBA-MenC ≥1:8, D42: number analyzed (Participants) | 346 | 341 | 116 | 687
  hSBA-MenC ≥1:8, D42 | 339 | 336 | 95 | 675
  hSBA-MenW-135 ≥1:4, D0: number analyzed (Participants) | 353 | 357 | 123 | 710
  hSBA-MenW-135 ≥1:4, D0 | 4 | 3 | 0 | 7
  hSBA-MenW-135 ≥1:4, D42: number analyzed (Participants) | 337 | 336 | 114 | 673
  hSBA-MenW-135 ≥1:4, D42 | 280 | 295 | 1 | 575
  hSBA-MenW-135 ≥1:8, D0: number analyzed (Participants) | 353 | 357 | 123 | 710
  hSBA-MenW-135 ≥1:8, D0 | 4 | 2 | 0 | 6
  hSBA-MenW-135 ≥1:8, D42: number analyzed (Participants) | 337 | 336 | 114 | 673
  hSBA-MenW-135 ≥1:8, D42 | 279 | 294 | 1 | 573
  hSBA-MenY ≥1:4, D0: number analyzed (Participants) | 344 | 349 | 122 | 693
  hSBA-MenY ≥1:4, D0 | 4 | 5 | 1 | 9
  hSBA-MenY ≥1:4, D42: number analyzed (Participants) | 333 | 329 | 117 | 662
  hSBA-MenY ≥1:4, D42 | 273 | 261 | 2 | 534
  hSBA-MenY ≥1:8, D0: number analyzed (Participants) | 344 | 349 | 122 | 693
  hSBA-MenY ≥1:8, D0 | 4 | 5 | 1 | 9
  hSBA-MenY ≥1:8, D42: number analyzed (Participants) | 333 | 329 | 117 | 662
  hSBA-MenY ≥1:8, D42 | 271 | 261 | 2 | 532

11. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers
Description: Anti-hSBA antibody titers were expressed as geometric mean titers (GMTs) for Nimenrix + Priorix-Tetra group, Nimenrix group, Meningitec group and Pooled group (Nimenrix + Priorix-Tetra and Nimenrix groups), respectively. The analysis was performed only on subjects receiving meningitis vaccination (Nimenrix) at Day 0.
Time Frame: Prior to first vaccine dose (Day 0) and 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Meningitec Group | Pooled Group
Number analyzed (Participants) | 359 | 363 | 123 | 722
Titer
  hSBA- MenA, D0: number analyzed (Participants) | 357 | 356 | 122 | 713
  hSBA- MenA, D0 | 2.1 [2.1 to 2.2] | 2.1 [2 to 2.1] | 2 [2 to 2.1] | 2.1 [2.1 to 2.2]
  hSBA- MenA, D42: number analyzed (Participants) | 348 | 338 | 117 | 686
  hSBA- MenA, D42 | 33.7 [28.9 to 39.2] | 19 [16.4 to 22.1] | 2 [2 to 2.1] | 25.4 [22.8 to 28.4]
  hSBA-MenC, D0: number analyzed (Participants) | 359 | 363 | 122 | 722
  hSBA-MenC, D0 | 2 [2 to 2] | 2 [2 to 2.1] | 2 [2 to 2.1] | 2 [2 to 2.1]
  hSBA-MenC, D42: number analyzed (Participants) | 346 | 341 | 116 | 687
  hSBA-MenC, D42 | 209.1 [183.8 to 238] | 196 [175.4 to 219] | 40.3 [29.5 to 55.1] | 202.5 [186 to 220.5]
  hSBA-MenW-135, D0: number analyzed (Participants) | 353 | 357 | 123 | 710
  hSBA-MenW-135, D0 | 2.1 [2 to 2.1] | 2.1 [2 to 2.1] | 2 [2 to 2] | 2.1 [2 to 2.1]
  hSBA-MenW-135, D42: number analyzed (Participants) | 337 | 336 | 114 | 673
  hSBA-MenW-135, D42 | 57.3 [47 to 69.9] | 48.9 [41.2 to 58] | 2 [2 to 2.2] | 52.9 [46.4 to 60.3]
  hSBA-MenY, D0: number analyzed (Participants) | 344 | 349 | 122 | 693
  hSBA-MenY, D0 | 2.1 [2 to 2.1] | 2.1 [2 to 2.1] | 2.1 [1.9 to 2.2] | 2.1 [2 to 2.1]
  hSBA-MenY, D42: number analyzed (Participants) | 333 | 329 | 117 | 662
  hSBA-MenY, D42 | 38.7 [32.2 to 46.7] | 30.9 [25.8 to 37.1] | 2.1 [1.9 to 2.3] | 34.6 [30.4 to 39.4]

12. Secondary Outcome: Anti-measles Antibody Concentrations
Description: Anti-measles antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL) in all groups.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 361 | 354 | 118 | 120
mIU/mL | 4273.4 [4018.4 to 4544.6] | 75 [75 to 75] | 4457.3 [3976.3 to 4996.6] | 75 [75 to 75]

13. Secondary Outcome: Anti-measles Antibody Concentrations
Description: Anti-measles antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in mIU/mL in a subset (30%) of the Nimenrix + Priorix-Tetra and Priorix-Tetra groups only. The analysis was performed only on subjects receiving varicella vaccination (Priorix-Tetra) at Day 0.
Time Frame: 42 days after the second Priorix-Tetra vaccine dose (Day 126)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Priorix-Tetra Group
Number analyzed (Participants) | 37 | 7
mIU/mL | 7113.8 [5335.6 to 9484.7] | 8699.8 [4865.3 to 15556.2]

14. Secondary Outcome: Anti-mumps Antibody Concentrations
Description: Anti-mumps antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in units per milliliter (U/mL) in all groups.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 349 | 354 | 116 | 120
U/mL | 662.9 [598.4 to 734.4] | 115.5 [115.5 to 115.5] | 710.1 [583.8 to 863.8] | 115.5 [115.5 to 115.5]

15. Secondary Outcome: Anti-mumps Antibody Concentrations
Description: Anti-mumps antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in U/mL in a subset (30%) of the Nimenrix + Priorix-Tetra and Priorix-Tetra groups only. The analysis was performed only on subjects receiving varicella vaccination ( Priorix-Tetra) at Day 0.
Time Frame: 42 days after the second Priorix-Tetra vaccine dose (Day 126)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Priorix-Tetra Group
Number analyzed (Participants) | 37 | 7
U/mL | 3351.2 [2658.2 to 4224.7] | 3334.1 [1933.1 to 5750.5]

16. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Anti-rubella antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in international units per millilier (IU/mL) in all groups.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 361 | 354 | 118 | 120
IU/mL | 43.1 [40 to 46.5] | 2 [2 to 2] | 53.2 [46.6 to 60.7] | 2 [2 to 2.1]

17. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Anti-rubella antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in IU/mL in a subset (30%) of the Nimenrix + Priorix-Tetra and Priorix-Tetra groups only. The analysis was performed only on subjects receiving varicella vaccination (Priorix-Tetra) at Day 0.
Time Frame: 42 days after the second Priorix-Tetra vaccine dose (Day 126)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Priorix-Tetra Group | Priorix-Tetra Group
Number analyzed (Participants) | 37 | 7
IU/mL | 87.2 [74.8 to 101.6] | 117 [73.8 to 185.5]

18. Secondary Outcome: Anti-varicella Antibody Titers
Description: Anti-varicella antibody titers were given as geometric mean titers (GMTs) for all groups.
Time Frame: 42 days after the first vaccine dose (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 333 | 335 | 111 | 116
Titers | 152.8 [133.5 to 174.8] | 2.2 [2 to 2.3] | 128.8 [99.1 to 167.4] | 2.2 [1.9 to 2.5]

19. Secondary Outcome: Anti-varicella Antibody Titers
Description: Anti-varicella antibody titers were given as geometric mean titers (GMTs) in a subset (30%) of the Nimenrix + Priorix-Tetra and Priorix-Tetra groups only. The analysis was performed only on subjects receiving varicella vaccination ( Priorix-Tetra) at Day 0.
Time Frame: 42 days after the second Priorix-Tetra vaccine dose (Day 126)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Priorix-Tetra Group | Priorix-Tetra Group
Number analyzed (Participants) | 36 | 7
Titers | 4175.6 [3064 to 5690.6] | 3360.1 [1646.5 to 6857]

20. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms Specific for Priorix-Tetra Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling for the Nimenrix + Priorix-Tetra Group and Priorix-Tetra Group, respectively. The analysis was performed only on subjects receiving varicella vaccination (Priorix-Tetra) at Day 0.
Time Frame: During the 4-day (Days 0-3) after vaccination with first dose of Priorix-Tetra vaccine at Day 0
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Priorix-Tetra Group
Number analyzed (Participants) | 375 | 124
Participants
  Pain | 75 | 22
  Redness | 126 | 48
  Swelling | 28 | 7

21. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms After Nimenrix or Meningitec Vaccination at Day 0
Description: Solicited local symptoms assessed were pain, redness and swelling for the Nimenrix + Priorix-Tetra Group, Nimenrix Group and Meningitec Group, respectively. The analysis was performed only on subjects receiving meningitis vaccination (Priorix-Tetra) at Day 0.
Time Frame: During the 4-day (Days 0-3) after vaccination with Nimenrix or Meningitec at Day 0
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Meningitec Group
Number analyzed (Participants) | 375 | 367 | 123
Participants
  Pain | 91 | 107 | 31
  Redness | 133 | 136 | 39
  Swelling | 52 | 69 | 10

22. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, fever (measured rectally and temperature ≥ 38.0°C ), irritability and loss of appetite, Meningismus, Parotiditis and Rash.
Time Frame: During the 4-day (Days 0-3) follow-up period after first vaccination dose in all groups
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 367 | 124 | 124
Participants
  Drowsiness | 122 | 103 | 29 | 40
  Fever≥38.0˚C | 56 | 34 | 14 | 16
  Irritability | 190 | 150 | 48 | 54
  Loss of appetite | 107 | 84 | 29 | 33
  Meningismus | 0 | 0 | 0 | 0
  Parotiditis | 0 | 0 | 0 | 0
  Rash | 22 | 23 | 10 | 6

23. Secondary Outcome: Number of Subjects With Priorix-Tetra - Specific Solicited General Symptoms
Description: Solicited general symptoms assessed were fever (measured rectally and temperature ≥ 38.0°C ), Meningismus, Parotiditis and Rash.
Time Frame: During the 43-day (Days 0-42) after first vaccination dose
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 367 | 124 | 124
Participants
  Fever ≥ 38.0˚C | 295 | 164 | 99 | 56
  Meningismus | 1 | 0 | 0 | 1
  Parotiditis | 0 | 0 | 0 | 0
  Rash | 119 | 66 | 36 | 24

24. Secondary Outcome: Number of Subjects Reporting Specific Adverse Events (AEs)
Description: Specific AEs include: rash, New Onset of Chronic Illness(es) (NOCI), and/or conditions prompting emergency room (ER) visits or non-routine physician office visits.
Time Frame: From Day 0 up to Month 6 after first vaccine dose
Population: The analysis was performed on the Total Vaccinated Cohort (TVC ), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 374 | 126 | 125
Participants
  Rash (es) | 13 | 10 | 2 | 6
  NOCI (s) | 6 | 3 | 1 | 1
  ER visit (s) | 28 | 29 | 3 | 7

25. Secondary Outcome: Number of Subjects Reporting Unsolicited Symptoms
Description: Unsolicited symptom covers any symptom reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 43-day (Days 0-42) post Dose 1 vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 374 | 126 | 125
Participants | 243 | 225 | 86 | 68

26. Secondary Outcome: Number of Subjects Reporting Unsolicited Symptoms
Description: as for outcome 25
Time Frame: During the 43-day (Days 0-42) follow-up period after each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 374 | 126 | 125
Participants | 252 | 233 | 90 | 75

27. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization, result in disability/ incapacity or are a congenital anomaly/ birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 6 after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Priorix-Tetra Group | Nimenrix Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 375 | 374 | 126 | 125
Participants | 13 | 10 | 3 | 2

ADVERSE EVENTS:
Time Frame: SAEs: Day 0 up to Month 6. Solicited local and general symptoms: 4-day after vaccination (Day 0-Day 3). Unsolicited symptoms: 43-day after vaccination (Days 0-42).
Description: The solicited local and general symptoms were only collected for those subjects who filled-in their symptom sheets.
Groups:
- Priorix-Tetra Group: Subjects received 1 dose of Priorix-Tetra™ vaccine on Day 0, one dose of Meningitec™ vaccine on Day 42 and a second dose of Priorix-Tetra™ vaccine on Day 84.
Arm/Group | Nimenrix + Priorix-Tetra Group | Meningitec Group | Nimenrix Group | Priorix-Tetra Group
All-Cause Mortality (participants affected / at risk) | 0/375 | 0/125 | 0/374 | 0/126
Serious Adverse Events (participants affected / at risk) | 13/375 | 2/125 | 10/374 | 3/126
Other Adverse Events (participants affected / at risk) | 340/375 | 103/125 | 313/374 | 108/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix + Priorix-Tetra Group (N=375) | Meningitec Group (N=125) | Nimenrix Group (N=374) | Priorix-Tetra Group (N=126)
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Medical observation (Investigations) | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1 | 0
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix + Priorix-Tetra Group (N=375) | Meningitec Group (N=125) | Nimenrix Group (N=374) | Priorix-Tetra Group (N=126)
Somnolence (Nervous system disorders) | 128 | 40 | 104 | 30
Irritability (Psychiatric disorders) | 210 | 56 | 161 | 58
Diarrhoea (Gastrointestinal disorders) | 53 | 16 | 40 | 14
Teething (Gastrointestinal disorders) | 39 | 13 | 38 | 14
Rhinitis (Infections and infestations) | 54 | 23 | 66 | 21
Upper respiratory tract infection (Infections and infestations) | 38 | 11 | 36 | 16
Otitis media (Infections and infestations) | 26 | 8 | 29 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 6 | 23 | 7
Decrease appetite (Metabolism and nutrition disorders) | 121 | 34 | 85 | 36
Erythema (Skin and subcutaneous tissue disorders) | 171 | 39 | 136 | 48
Pain (General disorders) | 112 | 31 | 111 | 22
Swelling (General disorders) | 66 | 10 | 70 | 7
Vomiting (Gastrointestinal disorders) | 20 | 2 | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.